CLINICAL TRIAL: NCT04497480
Title: Motor-Assisted and Active Resistive Upper/Lower Extremities Rehabilitation System for Treating Sarcopenia in Hospitalized Patients Aged 80 Years and Older
Brief Title: The Extremities Rehabilitation Training System for Sarcopenic Hospitalized Aged 80+ Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuxiang Liang (Other)
Responsible Party: Sponsor-Investigator, Yuxiang Liang, Physiotherapist, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020（001）
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Behavioral: Motor-Assisted and Active Resistive Upper/Lower Extremities Rehabilitation Training System
- controlled group (No Intervention)

INTERVENTIONS:
Behavioral: Motor-Assisted and Active Resistive Upper/Lower Extremities Rehabilitation Training System — The Passive, Motor-Assisted and Active Resistive Upper/Lower Extremities Rehabilitation Training System is designed for patients conﬁned to bed at the long-term care facilities hospitals, in early rehabilitation. This system can induce a natural movements of the upper/lower limb with safe motorized passive movement, as well as motor-assisted and active resistive muscle training to stimulate nerves, increase blood circulation of aﬀected tissue, cell metabolism and improve joint mobility, in promoting upper/lower extremities motor recovery.
  Arms: experimental group

SUMMARY:
Most previous clinical trials that addressed the rehabilitation training system for sarcopenic elderly subjects focused on community-dwelling older adults who were relatively healthy. There is a notable paucity of high-quality research investigating the effects and feasibility of the device for hospitalized or institutionalized older people, who are generally frailer and more severe in functional impairment than those living in the community. Moreover, most reported the system were of long-term duration, which typically lasted 3 to 6 months with two sessions per week. It remains unclear whether short-term the device training would be effective for treating sarcopenia. Therefore, the investigators aimed to assess the effectiveness of Motor-Assisted and Active Resistive Upper/Lower Extremities Rehabilitation Training System for treating sarcopenia in hospitalized older patients aged 80 years and over.

ELIGIBILITY:
Inclusion Criteria:

* Sarcopenia defined by the Asia Working Group of Sarcopenia (AWGS)
* Agree to participant this study and sign the informed consent
* Aged 80 years or over

Exclusion Criteria:

* Patients who could not follow the training plan due to cognitive impairment, emotional problems or any other reasons;
* Severe heart and lung diseases;
* Renal insufficiency;
* Any type of tumor;
* Bedridden patients

Ages: 80 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The change of activities of daily living | 3 Months
  Basic activities of daily living (BADL) assessed by Barthel Index

SECONDARY OUTCOMES:
The change of handgrip strength | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China